CLINICAL TRIAL: NCT01646463
Title: Integrative Stress Reduction for Maternal-Child Health
Brief Title: Pilot Trial of CenteringPregnancy With Mindfulness Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K01AT005270 (NIH)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Premature Birth; Low Birth Weight; Postpartum Depression
Keywords: mindfulness; stress; coping; emotion; depression; group medical visits; prenatal healthcare; preterm birth; birth weight; postpartum depression; cortisol; neuroendocrine function; blood pressure; health disparities
MeSH Terms: conditions — Premature Birth; Depression, Postpartum; Depression; Birth Weight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CenteringPregnancy with Mindfulness Skills (Experimental): CenteringPregnancy with Mindfulness Skills is the standard CenteringPregnancy prenatal healthcare intervention combined with mindfulness meditation and mindful movement/yoga applied to pregnancy, childbirth, and parenting.
  Interventions: Behavioral: CenteringPregnancy; Behavioral: CenteringPregnancy with Mindfulness Skills
- CenteringPregnancy (Active Comparator): CenteringPregnancy is group-based prenatal healthcare delivered according to the guidelines of the American College of Obstetrics and Gynecology. It includes assessment, support, and health education delivered in a healthcare empowerment framework.
  Interventions: Behavioral: CenteringPregnancy

INTERVENTIONS:
Behavioral: CenteringPregnancy — CenteringPregnancy (CP) follows a standardized curriculum for group-based prenatal healthcare offered to groups of 10-12 women with similar due dates. In lieu of receiving a series of individually-delivered prenatal healthcare, participants meet 10 times over the course of pregnancy and early postpartum for 2 hour sessions, essentially pooling their minutes for each prenatal healthcare visit. The visit schedule adheres to the guidelines set forth by ACOG of monthly and then weekly visits close to birth. All sessions of CP include three core components of: (1) physical assessment (including blood pressure, weight, and fundal height assessment), (2) education and skills-building, and (3) support. Content topics for group discussion include nutrition, exercise, relaxation, understanding pregnancy problems, infant care and feeding, postpartum issues including contraception, comfort measures in pregnancy, sexuality and childbearing, abuse issues, parenting, and childbirth preparation.
Behavioral: CenteringPregnancy with Mindfulness Skills — CenteringPregnancy with Mindfulness Skills contains the CenteringPregnancy (CP) content combined with training in mindfulness meditation and mindful movement/yoga. The mind-body methods have been adapted from those taught in the Mindfulness-Based Childbirth and Parenting (MBCP) course, which is a tailored version of the Mindfulness-Based Stress Reduction program delivered to pregnant women during the perinatal period. These practices include mindfulness meditation of the breath, body, feelings, thoughts, and emotions; body scan meditation; yoga postures practiced with mindful awareness of the body and the physical changes associated with pregnancy; and loving-kindness meditation. In addition, MBCP includes specific exercises in coping with stress, pain, and fear associated with pregnancy, childbirth, and early parenting with a focus on shifting the way participants relate to negative thoughts and emotions and cope with stress.
  Arms: CenteringPregnancy with Mindfulness Skills

SUMMARY:
In the U.S., rates of preterm birth and low birth weight have increased over the past 30 years. Poor birth outcomes are especially high among racial/ethnic minority populations. Maternal stress is an important factor that can lead to negative birth outcomes. Thus, programs that reduce stress during pregnancy could improve birth outcomes. Initial pilot work tested a mindfulness-based approach to stress reduction during pregnancy. Women in the pilot study had lower stress and improved coping after the program. For the current study, mindfulness is added to an existing prenatal healthcare program called CenteringPregnancy (CP). CP provides prenatal care through 10 group sessions. This study compares CP with a version of CP infused with mindfulness skills training. Effects of the two versions of CP on psychological stress and coping, stress hormones, and birth outcomes will be tested. Data will be collected from participants three times: twice during pregnancy and once after birth. Medical records will provide data on birth outcomes and other health factors. The study will provide initial information about a mind-body program to reduce stress and improve birth outcomes. Data from the study will inform the development of an R01 proposal for a larger study. The study will also help advance the long term goal of reducing health disparities.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and over
* enrolled to receive group-based prenatal healthcare from the San Francisco General Hospital (SFGH) Outpatient Midwifery Clinic CenteringPregnancy program

Exclusion Criteria:

* ineligible for CenteringPregnancy due to the need for individualized prenatal care
* Type 2 diabetes
* HIV
* seizure disorder
* serious mental health disorder
* substance abuse or medical condition that would lead to inability to adhere to intervention guidelines
* not fluent in English or Spanish
* previous formal training in meditation, yoga, or other mind-body practice
* previous participation in CenteringPregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-01; Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
preterm birth | post-birth
  gestational age at birth and risk of preterm birth (<37 weeks)
birth weight | post-birth
  birth weight in grams, birth weight to gestational age ratio, and risk of low birth weight (<2500 grams)
postpartum depression | post-birth
  incidence of self-reported postpartum depression

SECONDARY OUTCOMES:
change in and level of perceived stress | second trimester, third trimester, post-birth
  self-report of perceived life stress
change in and type(s) of coping | second trimester, third trimester, post-birth
  self-report of coping with salient stressful aspects of pregnancy and parenting
change in and level of mindfulness | second trimester, third trimester, post-birth
  self-report of mindfulness of daily experiences
change in and level of positive and negative emotion | second trimester, third trimester, post-birth
  self-report of intensity and frequency of positive and negative affect
change in and level of pregnancy-related anxiety | second trimester, third trimester
  self-report of pregnancy-related anxiety
change in and level of depressive mood | second trimester, third trimester
  self-report of depressive mood
change in and levels of salivary cortisol | second trimester, third trimester
  waking, 30-minutes post-waking, and bed-time salivary cortisol
change in and level of adrenocorticotropic hormone (ACTH) | second trimester, third trimester
  adrenocorticotropic hormone (ACTH) assayed from blood plasma
change in and levels of corticotropin releasing hormone (CRH) | second trimester, third trimester
  corticotropin releasing hormone (CRH) assayed from blood plasma
change in and levels of blood pressure | second trimester, third trimester
  diastolic and systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Larissa G Duncan, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States